CLINICAL TRIAL: NCT01924936
Title: Pilot Study of Online Interventions for Population-based Suicide
Brief Title: Now Matters Now: An Online Suicide Prevention Program
Acronym: NMN_SSIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Double | Purpose: Prevention
Other Study IDs: 1R34MH097836-01 (NIH); 1R34MH097836-01 (NIH)
Record Dates: First submitted 2013-07-17; First posted 2013-08-19 (Estimated); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Suicide; Suicide, Attempted; Suicidal Ideation
MeSH Terms: conditions — Suicide; Suicide, Attempted; Suicidal Ideation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Email (Placebo Comparator): Caring email (based on the caring letters literature) sent via secure email messaging. Of the interventions, it is by far the most minimal in clinical intensity and human resources needs for delivery.
  Interventions: Behavioral: DBT Online Program
- DBT program (Experimental): DBT online program involving three DBT skills taught across three lessons. The DBT online program will be based on a brief DBT skills intervention previously developed and pilot tested by Dr. Whiteside. This DBT online program will provide far greater clinical intensity than Intervention 1 and will be delivered with a widely-used modular software platform suitable for an R-34 project.
  Interventions: Behavioral: DBT Online Program
- Email + DBT program & Coach (Experimental): Caring Email + DBT online program & Coach: in addition to the DBT online program, will include personalized outreach and support for use of the program. An intervention "coach" will deliver this support exclusively via secure email messaging. The intervention coach will not provide psychotherapy, but instead provide reinforcement and contingency management surrounding completion of the three lessons. This intervention will utilize significantly greater ongoing clinical resources for its maintenance and offer greater clinical intensity for patients.
  Interventions: Behavioral: DBT Online Program

INTERVENTIONS:
Behavioral: DBT Online Program — DBT online program involving three DBT skills taught across three lessons. The DBT online program will be based on a brief DBT skills intervention previously developed and pilot tested by Dr. Whiteside. This DBT online program will provide far greater clinical intensity than Intervention 1 and will be delivered with a widely-used modular software platform suitable for an R-34 project.

SUMMARY:
In the United States in 2010, 38,000 people died from suicide and it is our nation's 10 leading cause of death. Suicide prevention is a national priority and yet secondary prevention programs targeting those most at risk are lacking. The purpose of the current research is to develop and pilot test three promising suicide prevention programs that, if found acceptable to high-risk individuals, could be further evaluated and eventually offered broadly and affordably to the public.

DETAILED DESCRIPTION:
Reducing the risk of suicide attempt and suicide is a public health priority. There has been no substantial decrease in suicide for the past two decades. Prevention efforts to date have focused on primary (e.g. public service announcements) and tertiary (e.g. interventions following suicide attempt) methods. Secondary or indicated prevention has been relatively unexplored. Secondary prevention requires both accurate screening methods and effective interventions. These essential elements are now available. Our recent research demonstrates that responses to the suicidal ideation item of the PHQ depression scale are a powerful predictor of subsequent suicide attempt and death. Availability of the PHQ in electronic medical records creates an opportunity for accurate population-level screening. Dialectical behavior therapy (DBT) has strong evidence of tertiary efficacy for preventing suicide attempts in clinical populations. Brief outreach tertiary interventions such as caring messages have some evidence for preventing suicide attempts. These clinical or tertiary prevention interventions provide the best available evidence for use in building secondary prevention programs. Resulting programs could then be linked to population-level screening data in electronic medical records. The first goal of the research plan is to adapt DBT and caring messages to fit delivery models suitable for the large numbers of at-risk patients identifiable in healthcare settings. The second goal is to evaluate the feasibility, acceptability, and safety of these alternative online suicide and self-injury secondary prevention programs. Online delivery models are suitable because they are scalable and can be provided securely, cheaply, and utilizing existing systems in healthcare. Three brief online interventions will be evaluated: caring email (CE); CE + DBT online program; and CE + DBT online program + coach. Each intervention will supplement usual care among high- risk patients identified via PHQ depression scales collected at outpatient primary care and mental health visits. Intervention content will be drawn from the principles of DBT and caring messages. The study design will be additive in order to examine alternative intervention models that vary widely in resources required for large- scale delivery. However, these interventions will require vastly fewer resources than in-person or telephone interventions. The project will involve intervention feasibility (pretesting, N=60) and acceptability and safety testing (pilot, N=400). Acceptability wll be assessed by patient intervention engagement levels (requiring the large pilot sample) and qualitative/formative intervention feedback from patients. Safety will be assessed via rates of psychiatric hospitalizations and self-injury diagnoses in the medical record in the intervention conditions compared to those receiving just continued usual care. Results of the pilot study will inform the design of a full-scale effectiveness trial examining the impact of one or more of these interventions on risk of suicide attempt and/or suicide death.

ELIGIBILITY:
Inclusion Criteria:

1. Group Health members who are ID verified for secure email messaging
2. Age 18 or older
3. Results of PHQ assessment completed with a medical provider (Group Health primary care or mental health) as part of ongoing care indicate increased risk for self-injury (item 9, 2 or 3 response)

Exclusion Criteria:

1. Patient has had a recent self-injury (past 60 days), as a more traditional clinical intervention would be more appropriate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2012-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Benchmark Acceptatiblity Rate | One Year
  For each intervention, we define one or more specific acceptability measures. These measures will be assessed using data from the electronic medical record and/or the intervention website. For each measure, we define a benchmark acceptability rate that we believe is necessary to proceed to further evaluation in a full-scale effectiveness trial. As discussed below, the proposed sample size will allow us to estimate these acceptability rates with confidence limits of approximately +/-9%. Consequently, we will establish "observed" benchmark rates that account for this level of precision. We do not propose to compare acceptability rates across intervention groups. Our objective is not comparison but description: to assess whether the observed acceptability rate for each intervention exceeds our threshold for proceeding to a full-scale evaluation.

SECONDARY OUTCOMES:
Number of Adverse Events | One Year
  Electronic medical records will be used to ascertain all suicide attempts and all psychiatric hospitalizations in each of the three intervention groups. Chi-square statistic will be used to determine whether any observed difference in rates of adverse outcomes exceeds that expected by chance. In addition, each of these events will be reviewed by study investigators (Whiteside and Simon) to assess possible relationship to the intervention program.

CONTACTS AND LOCATIONS:
Locations (1):
- Group Health Research Institute, Seattle, Washington, United States

REFERENCES:
- [Result] Whiteside U, Richards J, Simon GE. Brief Interventions via Electronic Health Record Messaging for Population-Based Suicide Prevention: Mixed Methods Pilot Study. JMIR Form Res. 2021 Apr 12;5(4):e21127. doi: 10.2196/21127. PMID 33843599
- See also: Related Info — https://formative.jmir.org/2021/4/e21127